CLINICAL TRIAL: NCT04461405
Title: INTEGRATE-D: A Pilot Test of Implementation Strategies to Support Integration of Medical and Psychosocial Care for People With Type II Diabetes
Brief Title: INTEGRATE-D: A Pilot Test to Support Integration of Medical and Psychosocial Care for People With Type II Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Deborah Cohen, Vice Chair for Research, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 20783; 5R34DK124146 (NIH)
Record Dates: First submitted 2020-06-26; First posted 2020-07-08 (Actual); Results first posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Type II Diabetes; Primary Health Care; Behavioral Health
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): INTEGRATE-D is a step-by-step blueprint that will assist practices with employing American Diabetes Association recommendations for integrating medical and psychosocial care. INTEGRATE-D consists of a set of implementation strategies that enable clinical teams to put evidence-based care in place. The intervention consists of training and education; audit and feedback materials; a facilitation implementation protocol; and health information technology support materials.
  Interventions: Behavioral: INTEGRATE-D
- Control Arm (No Intervention): Usual care

INTERVENTIONS:
Behavioral: INTEGRATE-D — INTEGRATE-D provides primary care practices with evidence-based training and support which includes: (1) Electronic health record (EHR)-based support-to help align EHR use with ADA recommendations and enable screening for depression, anxiety, DM distress, cognitive impairment, and self-management, and support identifying and tracking progress on patient treatments and goals; (2) Audit and feedback which involves assisting practices in accessing clinically relevant, actionable data reports to inform measurement and identification of care gaps in DMII and behavioral health care; (3) Skill-building resources including training on ADA-recommended care; and (4) Facilitation-to help implement the above strategies and the practice changes needed to align care with ADA recommendations.
  Arms: Intervention Arm

SUMMARY:
In 2016, the American Diabetes Association (ADA) published its first-ever recommendations for integrating medical and psychosocial care for patients with Type II Diabetes Mellitus (DMII) and common mental and behavioral health (MH/BH) problems. In the United States, 30 million people live with DMII, and the majority receive care in primary care settings. By implementing the ADA recommendations, primary care practices will help patients better manage their MH/BH needs, meet recommended goals for DMII management, and reduce the risk of adverse outcomes. Making these recommendations a routine part of practice is a major change, and it is critical to understand how best to implement the ADA recommendations and test its effectiveness in the real world. The pilot study builds on a series of prior studies to refine and pilot test a package of implementation strategies - called INTEGRATE-D - to support practices in implementing the ADA recommendations for integrated DMII care. INTEGRATE-D combines the following evidence-based implementation strategies: (1) electronic health record (EHR)-based support - to help align EHR use with ADA recommendations and enable screening for depression, anxiety, diabetes distress, cognitive impairment, and self-management, and support identifying and tracking progress on patient treatments and goals; (2) Audit and feedback - which involves assisting practices in accessing clinically relevant, actionable data reports to inform measurement and identification of care gaps in DMII and behavioral health care; (3) Skill-building resources - including training on ADA-recommended care; and (4) Facilitation - to help implement the above strategies and tailor the intervention so that practice work on the subset of areas where practices are ready to change to align care with ADA recommendations. The study aims are Aim 1: Refine the INTEGRATE-D intervention by incorporating the preferences of stakeholders. In partnership with patients, primary care key stakeholders and experts, compile and refine the package of implementation strategies in the INTEGRATE-D intervention. Aim 2: Demonstrate feasibility, acceptability, and estimate cost. Conduct a mixed-method, pre-post pilot comparing two practices that receive the INTEGRATE-D intervention to two control practices that receive training materials only.

DETAILED DESCRIPTION:
The INTEGRATE-D intervention is designed to support primary care practices with implementing ADA recommendations for integrating medical and psychosocial care for patients with DMII. Primary care practices will be the recipients of this support. For practices, the intervention will be 15 months long. The first three months will be a "Readiness Phase" where the study team assesses practices' capacity at baseline and a facilitator works with intervention practices to address capacity issues (e.g., help the practice produce a quality report) that can be barriers during active implementation. Then, intervention practices receive 12 months of "Active Intervention" with the same facilitator to align care processes with ADA recommendations. Pilot study design: The study team will use a randomized, mixed-method, pre-post design for this pilot study. The goal of this randomized pilot design is to evaluate the feasibility of recruitment, randomization, retention, assessment procedures, implementation of the INTEGRATE-D intervention, and provide insights into the effect of this pilot intervention on practice-level outcomes. Practice Sample and eligibility criteria: The sample for this pilot is four primary care practices. Practices with more than 100 adult patients (≥18 years) with a diagnosis of DM (Type II; not gestational) are eligible. Practice Recruitment: Practices will be recruited from the ORPRN practice-based research network. ORPRN works with 279 primary care practices in the state of Oregon, including 51% that are rural and 42% clinician-owned practices. ORPRN recruiters will identify 50 potential practices and conduct a faxback to assess interest, capacity, and eligibility. Of interested practices, ORPRN and the study team will select 4 practices (2 rural and 2 non-rural) that vary on whether practices employ a behavioral health clinician. The study team will purposefully vary practices on these characteristics based on previous work that demonstrated they influenced intervention uptake. Patient Sample: The study team will have three different patient samples. For chart audits, there will be two samples. (1) Patients with a diagnosis of DMII who have been seen at least once at the practice in the 15 months prior to the intervention start date and at least once after the intervention start date will be included in the chart audit. The study team will randomly select 50 patients meeting these criteria. (2) Patients meeting the above criteria and screening positive for depression (i.e., those patients who have minimally exposed to the INTEGRATE-D intervention will also be randomly selected for chart audit. The study team will audit charts until there is a sample of 30 patients meeting these criteria. (3) From this latter group, the study team will select 5 patients at each of the two intervention practices to participate in an interview. Randomization Procedure: Practices will be randomized in a 1:1 ratio through a covariate-constrained randomization procedure. This is accomplished as follows. Prior to randomization, the study team will collect baseline data on practice-level factors (e.g., practice size, ownership, rurality, patient panel demographics, etc.) that could influence process and outcome measures. These data will be collected as part of the recruitment process. The study team will construct all possible combinations of eligible practices into two groups. For each selected possible randomization, the study team will compare the balance between study arms in the important baseline data described above through a balance criterion. The study team will randomly select one randomization combination (from the 2 combinations with the best balance) which will yield 2 practices in each study arm with good balance in important covariates. Data Collection: For this pilot study, the study team will collect mixed methods (survey, observation, interview, and chart audit) data. For control practices, data collection will include the collection of survey and chart audit data. These data will be collected at the same time as data collected from intervention practices. Intervention practices, in addition to completing surveys and participating in the chart audit, will participate in practice site visits, which include the study team observing the practice and how it delivers care and interviewing a varied group of practice members, including those that participated in implementing the intervention. These visits will happen before and after the intervention. In addition, during the implementation of INTEGRATE-D, the study team will conduct monthly telephone calls with a key informant at the intervention practices. Measures: The study team will measure practice capacity for quality improvement using the Change Process Capability Questionnaire (survey). The study team will measure changes in care processes, as follows: for depression - screening for depression using the Patient Health Questionnaire (PHQ)-9, rates of referral to behavioral health when patients screen positive on the PHQ-9; for diabetes - the study team will use a composite measure of DMII process of clinical care (e.g., screening for HbA1c, eye, and foot exams) and assess discussion of and engagement in self-management activities (e.g., healthy eating, physical activity). The study team will measure outcome change as a change in PHQ-9 and HbA1c. All process and outcome measures will all be collected via chart audit. The study team will measure feasibility and acceptability, perceived and actual, of INTEGRATE-D using observation, semi-structured interviews, survey, and facilitator tracking data. Surveys will use validated acceptability and feasibility measures. Statistical power: As this is a pilot study, it is not meant to have the sample size needed to test for statistical significance. Rather, this pilot is designed to show the promise of the INTEGRATE-D intervention and provide the data need to do accurate power calculations for the larger, subsequent pragmatic trial. Data Analysis. Qualitative analysis will follow a rigorous process whereby a team of experienced qualitative researchers will identify emerging patterns or findings, and then analyze data again to solidify these patterns into a coherent set of findings. Quantitative analyses will use standard descriptive statistical methods and the study team will utilize Generalized Linear Mixed Models to compare the effect of INTEGRATE-D intervention on process outcome measures in the context of a cluster-randomized design.

ELIGIBILITY:
Inclusion Criteria

In order for patients to become eligible, their primary care practice must meet the following inclusion criteria:

* Primary care practices are affiliated with the Oregon Rural Practice-Based Network (ORPRN), at time of recruitment.
* Primary care practices must be located in Oregon.
* Primary care practices have more than 100 adult patients aged 18 years or older with an electronic health record-based diagnosis of Type II Diabetes Melitus (DMII).

Once the criteria for a primary care practice is satisfied, the inclusion criteria for DMII patients includes the following:

* Patients are 18 years of age or older.
* Patients have an electronic health record-based diagnosis of DMII.
* Patients were seen by an ORPRN practice at least once in the 15 months prior to the start of intervention and once during the intervention.

Exclusion Criteria

Primary care practices that do not meet the inclusion criteria established are not eligible for the pilot study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 294 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Cohen, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited four clinics that varied on location, size, ownership, and specialty mix. Clinics were enrolled in March 2020. Data collection was completed in July 2022.
Pre-assignment Details: From each of the four recruited clinics, two samples of patients were randomly selected for chart abstraction: (1) 50 patients with a diagnosis of type 2 diabetes and (2) 30 patients with a diagnosis of type 2 diabetes and depression or Diabetes Distress (DD), with the exception of the second Intervention clinic, for which only 4 patients could be recruited for the second sample. Between Intervention and Control arms, a total of 294 patients were selected for chart abstraction.
Units Other Than Participants: Clinics
Period: Overall Study
Arm/Group | Intervention Arm | Control Arm
Started | 134; 2 Clinics | 160; 2 Clinics
Completed | 134; 2 Clinics | 160; 2 Clinics
Not Completed | 0; 0 Clinics | 0; 0 Clinics

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Arm | Control Arm | Total
Number analyzed (Participants) | 134 | 160 | 294
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 76 | 73 | 149
  >=65 years | 58 | 87 | 145
Age, Continuous [Mean (Standard Deviation); unit: years]
  mean (SD) | 60.28 (13.11) | 65.53 (13.41) | 63.14 (13.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 80 | 161
  Male | 53 | 80 | 133
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 10 | 33
  Not Hispanic or Latino | 100 | 141 | 241
  Unknown or Not Reported | 11 | 9 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 5 | 12 | 17
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
  Black or African American | 4 | 2 | 6
  White | 116 | 134 | 250
  More than one race | 3 | 0 | 3
  Unknown or Not Reported | 4 | 9 | 13
Region of Enrollment [Number; unit: participants]
  United States | 134 | 160 | 294
Hba1c [Mean (Standard Deviation); unit: percentage of Hba1c] | 7.50 (1.63) | 7.12 (1.34) | 7.30 (1.49)

OUTCOME MEASURES:

1. Primary Outcome: Acceptability of Intervention
Description: A post-intervention four-item survey that evaluates the extent to which the intervention meets practice members' approval, is appealing and is liked and welcomed. The items were assessed on a Likert scale, ranging from -2 to 2 (i.e., completely disagree to completely agree, with 0 indicating neutrality). Composite scores were created by averaging scores for the four individual items. The scale range is from -2 (minimum) to +2 (maximum), where higher values represent a better outcome (more approval).
Time Frame: At 15 months, post-intervention
Population: Practice members at intervention clinics.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Clinics
Groups:
- Intervention Clinics: A survey measuring the acceptability, appropriateness, and feasibility of the intervention was collected from clinic members exposed to the intervention.
Arm/Group | Intervention Clinics
Number analyzed (Participants) | 13
Number analyzed (Clinics) | 2
units on a scale | 0.60 (0.50)

2. Primary Outcome: Feasibility of the Intervention
Description: A post-intervention four-item survey that evaluates the extent to which the intervention is implementable, seems possible, seems doable, and seems easy to use. The items were assessed on a Likert scale, ranging from -2 to 2 (i.e., completely disagree to completely agree, with 0 indicating neutrality). Composite scores were created by averaging scores for the four individual items. The scale range is from -2 (minimum) to +2 (maximum), where higher values represent a better outcome (more approval).
Time Frame: At 15 months, post-intervention
Population: Practice members at intervention clinics
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Clinics
Arm/Group | Intervention Clinics
Number analyzed (Participants) | 13
Number analyzed (Clinics) | 2
units on a scale | 0.50 (0.43)

3. Primary Outcome: Appropriateness of Intervention
Description: as for outcome 1
Time Frame: At 15 months, post-intervention
Population: Practice members at intervention clinics
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Clinics
Arm/Group | Intervention Clinics
Number analyzed (Participants) | 13
Number analyzed (Clinics) | 2
units on a scale | 0.79 (0.45)

4. Secondary Outcome: Change in Hemoglobin A1c
Description: Difference between baseline and end-of-intervention average blood sugar levels.
Time Frame: Baseline (pre-intervention) and 15-months (post-intervention).
Measure: Mean (Standard Deviation); unit: percentage of Hba1c
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 134 | 160
percentage of Hba1c | -0.04 (1.56) | -0.08 (1.35)

5. Secondary Outcome: Change in Patient Health Questionnaire-9 (PHQ-9)
Description: Difference between baseline and end-of-intervention PHQ-9 score.
  PHQ-9: This nine-item validated screener measures depression severity. Questionnaire items are on a Likert scale and range from 0 (i.e., not at all) to +3 (i.e., nearly every day), and the total score ranges from 0 (i.e., minimal to none) to 27 (i.e., severe).
Time Frame: Baseline (pre-intervention) and 15-months (post-intervention).
Population: This outcome measure was only assessed among the sample of patients with a diagnosis of type 2 diabetes and depression or Diabetes Distress (DD).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 34 | 60
units on a scale | -1.25 (6.72) | 2.44 (6.69)

ADVERSE EVENTS:
Time Frame: Two years and four months (March 01, 2020 to July 01, 2022)
Description: Clinicians would inform our team if there was an adverse event.
Arm/Group | Intervention Arm | Control Arm
All-Cause Mortality (participants affected / at risk) | 0/134 | 0/160
Serious Adverse Events (participants affected / at risk) | 0/134 | 0/160
Other Adverse Events (participants affected / at risk) | 0/134 | 0/160

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-10-26): https://cdn.clinicaltrials.gov/large-docs/05/NCT04461405/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-26): https://cdn.clinicaltrials.gov/large-docs/05/NCT04461405/SAP_001.pdf